CLINICAL TRIAL: NCT02118142
Title: Modulation of Insulin Sensitivity by Betaine Upregulation of FGF21
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Nutrition Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 13-2548
Record Dates: First submitted 2014-04-02; First posted 2014-04-21 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance | interventions — Betaine; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Betaine (Active Comparator): 6 gram dose of betaine delivered in encapsulated form
  Interventions: Dietary Supplement: Betaine
- Dextrose (Placebo Comparator): 6 gram dose of dextrose delivered in encapsulated form
  Interventions: Dietary Supplement: Dextrose

INTERVENTIONS:
Dietary Supplement: Betaine — 6 gram one-time dose of betaine delivered in encapsulated form with an unsweetened beverage
  Arms: Betaine
Dietary Supplement: Dextrose — 6 gram one-time dose of dextrose delivered in encapsulated form with an unsweetened beverage
  Arms: Dextrose

SUMMARY:
People with poor insulin sensitivity do not respond normally to elevations in blood sugar. This may increase their risk of developing diabetes in the future. The purpose of this research study is to determine if the nutrient betaine, found in beets, spinach and wheat products, can enhance the production of fetal growth factor 21 (FGF21), a molecule that is believed to promote insulin sensitivity.

DETAILED DESCRIPTION:
AIM: To determine if betaine is a modulator of FGF21 in humans. Low plasma betaine is associated with an increased risk of metabolic syndrome, but the mechanisms modulating this correlation are poorly delineated. Betaine bioavailability in humans is determined by dietary intake and genetic polymorphisms that influence betaine metabolism. Therefore, moderating betaine levels could be particularly beneficial for some individuals. FGF21 is elevated in response to insulin insensitivity and is under active investigation as a therapeutic modality. The mechanisms of action of FGF21 and betaine on insulin sensitivity in humans are incompletely understood. This study tests the hypothesis that betaine induces FGF21 secretion and insulin sensitizing actions in humans by measuring plasma FGF21, betaine, choline (betaine precursor), glucose, insulin and adiponectin in response to betaine supplementation over a 24 hour time course in 20 healthy, lean individuals. This pilot nutrition intervention will provide key preliminary evidence for understanding whether and how betaine exerts metabolic benefit in humans and will inform a future study to investigate the novel betaine-FGF21-insulin sensitivity axis in a larger cohort.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Able/willing to consume study meals
* Non-smoker
* BMI in normal range (18-24.9)

Exclusion Criteria:

* Use of chronic medications
* Abnormal physical examination or chronic illness
* Use of drugs or medications known to alter choline/betaine metabolism
* Consumption of more than 2 oz of alcohol/day or 24 oz wine/day
* Use of choline/betaine-containing dietary supplements during the previous 3 months
* Diagnosed with Cystathionine Beta-Synthase (CBS) Deficiency
* Pregnant or breastfeeding
* Known hypersensitivity to betaine
* Current substance abuse or addiction

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Plasma Fetal Growth Factor 21 (FGF21) concentration | 0, 0.5, 1, 2, 4, 8, and 24 hours post- betaine or placebo supplement
Plasma choline concentration | 0, 0.5, 1, 2, 4, 8, and 24 hours post- betaine or placebo supplement
Plasma betaine concentration | 0, 0.5, 1, 2, 4, 8, and 24 hours post- betaine or placebo supplement
Plasma glucose concentration | 0, 0.5, 1, 2, 4, 8, and 24 hours post- betaine or placebo supplement
Plasma insulin concentration | 0, 0.5, 1, 2, 4, 8, and 24 hours post- betaine or placebo supplement
Plasma adiponectin concentration | 0, 0.5, 1, 2, 4, 8, and 24 hours post- betaine or placebo supplement

SECONDARY OUTCOMES:
Typical dietary intake | During day 2 of the first 3 day phase
  Assessed via questionnaire
Typical exercise habits | During day 2 of the first 3 day phase
  Assessed via questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Karen Corbin, PhD, RD, Principal Investigator — UNC Nutrition Research Institute
Locations (1):
- UNC Nutrition Research Institute, Kannapolis, North Carolina, United States